CLINICAL TRIAL: NCT01301846
Title: Participation of Manual Wheelchair Users in the Community: The Relationship to Wheelchair Skills Capacity
Brief Title: Participation of Manual Wheelchair Users in the Community
Status: Withdrawn | Type: Observational
Why Stopped: Need to recruit research staff
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Kim Parker, Rehabilitation Engineer, Nova Scotia Health Authority
Other Study IDs: CDHA-RS/2011-082
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Wheelchairs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Wheelchair users: People who have a wheelchair for home and community use.

SUMMARY:
To explore the relationship between ability to do different wheelchair skills and the participation and quality of life of wheelchair users in and around their home and community. The investigators study hypothesis:

1. Self-reported capacity of wheelchair skills (ability to do wheelchair skills) is strongly related to self-reported participation.
2. Self-reported capacity of wheelchair skills (ability to do wheelchair skills) is related to the average daily distance traveled in their wheelchair.

ELIGIBILITY:
Inclusion Criteria:

* have a manual wheelchair for home and community use;
* use a manual wheelchair at least once a week;
* have a minimum of 3 months experience using a manual wheelchair outside the hospital setting;
* be over the age of 18;
* be able to read and understand English and follow verbal and visual instructions;
* be competent to give informed consent;
* be willing to take part in the study, including signing the consent after carefully reading it;
* not have been under significant bed rest for the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of people who use manual wheelchairs
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Wheelchair Skills Test Questionnaire Capacity Version | baseline
  Participants will be asked if they can perform 32 skills from the WST 4.1 (capacity)using a structured interview approach. A skill will be considered a pass if done describing a safe manner.
Impact on Participation and Autonomy Questionnaire | baseline
  This measure addresses autonomy with respect to activities and participation, and is a self-report measure.
Average Distance Travelled | Up to a week time period, one time measure
  The average distance treavelled per day over a week in the participant's wheelchair will be measured.

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale short form | baseline
  Self-reported depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada